CLINICAL TRIAL: NCT06144645
Title: A Phase 3, Randomized, Double-Blind, Dose-Ranging Evaluation of Transcutaneous Vagus Nerve Stimulation (tVNS) to Reduce Temper Outbursts in People With Prader-Willi Syndrome (PWS)
Brief Title: A Clinical Evaluation of Non-Invasive Vagus Nerve Stimulation for Temper Outbursts in People With PWS
Acronym: VNS4PWS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Foundation for Prader-Willi Research (Other)
Collaborators: RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FPWR-VNS-R-3-01
Record Dates: First submitted 2023-10-16; First posted 2023-11-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; PWS; Prader
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tVNS, Intermittent Stimulation (Active Comparator): 28 seconds on, 32 seconds off
  Interventions: Device: tVNS, intermittent stimulation
- tVNS, Continuous Stimulation (Active Comparator): continuous stimulation
  Interventions: Device: tVNS, continuous stimulation

INTERVENTIONS:
Device: tVNS, intermittent stimulation — transcutaneous vagus nerve stimulation, intermittent stimulation
  Other Names: tVNS R, manufactured by tVNS Technologies, intermittent stimulation
  Arms: tVNS, Intermittent Stimulation
Device: tVNS, continuous stimulation — transcutaneous vagus nerve stimulation, continuous stimulation
  Other Names: tVNS R, manufactured by tVNS Technologies, continuous stimulation
  Arms: tVNS, Continuous Stimulation

SUMMARY:
The goal of the VNS4PWS clinical study is to test the efficacy, safety, and acceptability of transcutaneous vagus nerve stimulation (tVNS) treatment in people with PWS.

DETAILED DESCRIPTION:
The main questions the VNS4PWS study seeks to answer are: (1) is tVNS treatment safe in people with PWS, (2) is tVNS treatment acceptable to people with PWS, and (3) is tVNS an effective treatment to reduce temper outbursts in people with PWS. Participants will wear the tVNS device daily for 4 hours over a period of 9 months. Two different doses of tVNS will be compared. During the final three months of the trial, the effect of stopping treatment will be studied. After the first year of the study, participants will have the opportunity to continue on to a 1-year open label extension period during which active tVNS treatment will be resumed.

ELIGIBILITY:
Inclusion Criteria:

1. Genetically proven diagnosis of PWS.
2. Age 10-40 years.
3. History in the last six months of an average of at least two temper outbursts per week.
4. Able to comply with requirements of study and provide consent or assent; If consent is to be provided by the participant's guardian, same applies to the guardian.
5. Concomitant use of psychiatric medication is allowed; participant must be on a stable dose 90 days prior to screening with no plans for dose modification during the course of the study.
6. Concomitant use of psychotherapy/counseling is allowed. Therapies for mental health or behavior challenges, including applied behavior analysis (ABA) are also allowed; however, participant must be on a stable regimen 90 days prior to screening with no plans for modification during the course of the study.
7. Living with family or in another setting with family members or staff willing to support the participant and the required data collection.
8. Agree to share tVNS patient application compliance and daily temper outburst data with the sponsor.
9. Access to cellular data or Wi-Fi.
10. Participant and caregiver speak American English as first language or are fluent in American English.

Exclusion Criteria:

1. Positive pregnancy test at screening, baseline, or at any point in the study.
2. Evidence of active or recent unstable serious mental illness, including, psychosis, mania, severe depression, or suicidality.
3. Moved to present residential placement in last three months or less.
4. Likely move in residential placement during the course of the study.
5. Cardiac abnormalities including medically documented history of cardiac disease or cardiac arrhythmia, documented resting heart rate ≤ 50 beats per minute (BPM); or history of 2° type 2 or 3° heart block on electrocardiogram (ECG).
6. Evidence of clinically significant abnormalities of blood, liver, or kidney function from clinical safety laboratory assessments as determined by the Site Investigator.
7. History of blood clot, pulmonary embolism, or deep vein thrombosis.
8. Prior diagnosis of epilepsy or currently active seizures.
9. Current enrollment in the active phase of different clinical trial or interventional study.
10. Current use of hearing aids or implantable medical devices including implanted vagus nerve stimulation (iVNS) device, implanted cardiac pacemaker, implanted cardiac defibrillator, cochlear implants, cerebral shunt or cardiac implantable electrical devices.
11. Presence of dermal abnormalities at the stimulation site that would interfere with the ability of the tVNS device to function properly.
12. Presence of an allergy to titanium, titanium-iridium, thermoplastic elastomers, perfluoroethylene propylene, or polyurethane elastomers, or components of / preservatives present in the device electrode cream (Ceteareth-20, Propylene Glycol, Bentonite, Polysorbate 20, Phenoxyethanol, Ethylhexylglycerin).
13. Severe, untreated sleep apnea, as self-reported by subject or caregiver or suspected by Site Investigator.
14. Subject is, in the opinion of the Investigator, not suitable to participate in the study.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine the safety profile and tolerability of tVNS in PWS, as assessed by the frequency, severity, and seriousness of adverse events determined during the study. | Through study completion, an average of 1 year
  Frequency, severity, and seriousness of adverse events during the study.
To determine the acceptability profile of tVNS in PWS as assessed by the rate of withdrawal from the study. | Through study completion, an average of 1 year
  The acceptability profile of tVNS in PWS will be measured by the rate of withdrawal from the study.
To determine the acceptability profile of tVNS in PWS as assessed by the rates of device use compliance during the study. | Through study completion, an average of 1 year
  The acceptability profile of tVNS in PWS will be measured by the rates of device use compliance throughout the study.
To determine the efficacy of tVNS in reducing temper outbursts in people with PWS aged 10 - 40 years. | Baseline to month 9
  Change in Aberrant Behavior Checklist, irritability subscale. A lower score indicates a better outcome whereas a higher score indicates a worse outcome. The minimum score is zero and the maximum score is 45.

SECONDARY OUTCOMES:
To determine the efficacy of tVNS in reducing temper outbursts in people with PWS aged 10 - 40 years over the course of the study as assessed by the irritability subscale of the Aberrant Behavior Checklist. | Baseline to months 3, 6, 9.
  Aberrant Behavior Checklist irritability subscale. A lower score indicates a better outcome whereas a higher score indicates a worse outcome. The minimum score is zero and the maximum score is 45.
To determine whether tVNS reduces the average number of temper outbursts per day, as assessed by the Daily Survey. | Baseline to months 3, 6, 9, and 12.
  The Daily Survey will collect caregiver-reported data on the number of temper outbursts per day. A lower score indicates a better outcome and a higher score indicates a worse outcome. The minimum daily score is zero and the maximum daily score that the scale can capture is 20.
To determine whether tVNS reduces the average intensity of daily temper outbursts as measured by the Daily Survey. | Baseline to months 3, 6, 9, and 12.
  The Daily Survey will collect caregiver-reported data on the intensity of daily temper outbursts. A higher score indicates a worse outcome and a lower score indicates a better outcome. The minimum score is 1 and the maximum score is 7.
To determine whether tVNS reduces the average duration of temper outbursts per day. | Baseline to months 3, 6, 9, and 12.
  The Daily Survey will collect caregiver-reported data on the duration of daily temper outbursts. The minimum score is 1 and the maximum score is 7.
To determine whether tVNS decreases PWS-associated hyperphagic behaviors as measured by the Hyperphagia Questionnaire for Clinical Trials. | Baseline to months 3, 6, and 9.
  Stimulation of the vagus nerve may impact hyperphagic drive. It may also impact eating behaviors and the ability of the person with PWS to cope with eating restrictions. Higher scores indicate a worse outcome and lower scores indicate a better outcome. The minimum score is 0 and the maximum score is 36.
To determine whether tVNS treatment decreases skin picking in PWS, as assessed by the Self Injury Trauma Scale. | Baseline to months 3, 6, and 9.
  The Self Injury Trauma Scale is a widely used method for quantifying surface tissue damage caused by self-injurious behavior. A lower score indicates a better outcome and a higher score indicates a worse outcome. The minimum score is 1 and the maximum is 5.
To determine whether tVNS decreases anxiousness and distress in PWS as measured by the PWS Anxiousness and Distress Questionnaire. | Change in PWS Anxiousness and Distress Questionnaire at baseline and months 3, 6, and 9.
  tVNS may impact behaviors associated with anxiousness and distress, which are common in PWS. A lower score indicates a better outcome and a higher score indicates a worse outcome. The minimum score is 0 and the maximum is 56.
To determine whether reductions in temper outbursts result in reduced caregiver burden as measured by the Zarit Burden Interview. | Change in Zarit Burden Interview (ZBI) between baseline and month 9.
  Reduction in outbursts is expected to positively impact other members of the participant's family - this measure may reflect improvements in family relationships. A higher score indicates a worse outcome. A lower score indicates a better outcome. The minimum score is 0 and the maximum score is 88.
To determine whether reductions in temper outburst is associated with improved quality of life as measured by the Parent Proxy Global Health 7. | Change in Parent Proxy Global Health 7 from baseline to months 3, 6, 9.
  Reduction in outbursts is expected to meaningfully improve quality of life as assessed by the Parent Proxy Global Health 7. A higher score indicates a better outcome and a lower score indicates a worse outcome. The minimum score is 7. The maximum score is 35.
To assess whether overall disease severity is improved as measured by the Change in the Clinical Global Impression of disease severity. | Change in the Clinical Global Impression of disease severity at baseline and months 3, 6, 9.
  This measure will serve as an anchor to assess the meaningfulness of reductions in temper outbursts. A lower score indicates a better outcome. A higher score indicates a worse outcome. The maximum score is 7. The minimum score is 1.
To assess whether there is a global improvement in behavior as assessed by the Clinical Global Impression of Improvement. | Change in the Clinical Global Impression of Improvement from baseline to months 3, 6, 9.
  Global changes in behavior and will serve as an anchor to assess the meaningfulness of change. A lower score indicates a better outcome. A higher score indicates a worse outcome. The maximum score is 7. The minimum score is 1.

OTHER OUTCOMES:
Informant and self-reported measures of acceptability as assessed by a qualitative exit interview. | Through study completion, an average of 1 year.
  To qualitatively determine the acceptability of tVNS in people with PWS and to better understand specific reasons for discontinuation that occurred in this study.
Identification of responder characteristics as identified in a qualitative exit interview. | Through study completion, an average of 1 year.
  Participant characteristics and information provided in semi-structured exit interviews will inform efforts to identify those most likely to benefit from this intervention.
To assess the change heart rate variability (HRV) in a subset of participants. | Through study completion, an average of 1 year.
  Heart rate variability is abnormal in PWS, and VNS may cause changes in HRV.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Strong, PhD, Principal Investigator — Foundation for Prader-Willi Research; Deepan Singh, MD, Principal Investigator — Maimonides Medical Center
Locations (18):
- United States (18):
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Rare Disease Research, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Health, Garden City, New York
  - Montefiore Medical Center and Albert Einstein College of Medicine, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Christus Children'S, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No